CLINICAL TRIAL: NCT04852588
Title: Endoscopic Nodal Staging in Oligometastatic Non-small Cell Lung Cancer (NSCLC) Being Treated With Stereotactic Ablative Radiotherapy (ENDO-SABR)
Brief Title: Chest Lymph Node Sampling in Patients With Advanced Lung Cancer to be Treated With Curative-intent Radiation Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-SABR; ReDA #11162 (Other: Lawson Health Research Institute)
Record Dates: First submitted 2021-04-12; First posted 2021-04-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Oligometastatic Non-Small Cell Lung Cancer; Stereotactic Ablative Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Small pieces of suspicious chest lymph nodes will be removed with a procedure called endobronchial ultrasound-guided transbronchial fine needle aspiration (EBUS-TFNA) or transesophageal ultrasound-guided fine needle aspiration (EUS-FNA).
  Interventions: Procedure: Endobronchial ultrasound-guided transbronchial fine needle aspiration (EBUS-TFNA); Procedure: Transesophageal ultrasound-guided fine needle aspiration (EUS-FNA)

INTERVENTIONS:
Procedure: Endobronchial ultrasound-guided transbronchial fine needle aspiration (EBUS-TFNA) — Chest lymph node sampling procedure by EBUS
Procedure: Transesophageal ultrasound-guided fine needle aspiration (EUS-FNA) — Chest lymph node sampling procedure by EUS

SUMMARY:
This study will investigate the role of sampling suspicious chest lymph nodes with a procedure called endobronchial ultrasound-guided transbronchial fine needle aspiration (EBUS-TFNA) or transesophageal ultrasound-guided fine needle aspiration (EUS-FNA) in patients planned to receive radical dose radiation.

This study will use Stereotactic Ablative Radiotherapy (SABR) for treatment methods. SABR is a newer radiation treatment that delivers high-dose, precise radiation to small tumors and can be delivered more accurately than with older radiation treatment methods. It is considered a standard treatment for small lung cancers, and select cancers that have spread to the brain.

The purpose of this study is to compare if the lymph node sampling procedure is valuable for determining the extend of nodal disease in metastatic Non-Small Cell Lung Cancer (NSCLC) compared to imaging alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oligometastatic non-small cell lung cancer (NSCLC), including a primary lung tumour (± hilar/mediastinal adenopathy) with up to 5 synchronous metastases
* Radical treatment intent to all sites is recommended at multi-disciplinary tumour board or by discussion by medical oncologist and radiation oncologist and/or surgeon.
* Age 18 years or older
* Good performance status (Eastern Cooperative Oncology Group [ECOG 0-1) with life-expectancy of at least 6 months as determined by enrolling physician
* Patient has undergone staging investigations less than 3 months prior to registration.

  1. Positron Emission Tomography (PET) / Computed Tomography (CT) and Magnetic Resonance Imaging (MRI) brain (CT brain with contrast if contraindication to MRI) OR
  2. CT chest/abdomen, radionucleotide bone scan and MRI of brain (CT brain with contrast if contraindication to MRI)
* Pathologic confirmation of NSCLC

Exclusion Criteria:

* Contraindication to Endobronchial Ultrasound (EBUS) / Endoscopic Ultrasound (EUS)
* Unable to provide consent for EBUS/EUS
* Contraindication to chest radiotherapy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes to treatment intent and/or plan | 2 years
  Number of patients whose treatment is changed from stereotactic ablative radiotherapy (SABR) to conventional dose radiation, change in mediastinal radiation field, change from curative intent to palliative intent treatment

SECONDARY OUTCOMES:
Determine the proportion of patients with occult mediastinal metastasis | 2 years
  Pre-staging treatment planning anticipated lymph nodes to be treated compared to post staging lymph nodes to be treated
Determine the sensitivity and specificity of radiologic staging of hilar/mediastinal lymph nodes | 2 years
  Nodal staging on imaging alone versus nodal staging after sampling
Identify the total number of lymph nodes sampled per procedure | 2 years
  Record the total number of lymph nodes sampled
Identify the nodal stations sampled | 2 years
  Record the nodal stations that were sampled
Determine the proportion of patients with complications of endoscopic procedure | 2 years
  Number of participants with complications versus number without

CONTACTS AND LOCATIONS:
Overall Officials: Inderdeep Dhaliwal, MD, Principal Investigator — London Health Sciences Centre, Lawson Health Research Institute
Locations (2):
- Canada (2):
  - London Health Sciences Centre - London Regional Cancer Program, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhaliwal I, Kassirian S, Mitchell MA, Qiabi M, Warner A, Louie AV, Wong HH, McDonald CM, Rajchgot J, Palma DA. Endoscopic nodal staging in oligometastatic non-small cell lung cancer (NSCLC) being treated with stereotactic ablative radiotherapy (ENDO-SABR). BMC Cancer. 2022 Apr 28;22(1):468. doi: 10.1186/s12885-022-09563-8. PMID 35484614